CLINICAL TRIAL: NCT01568827
Title: Inflammation, Polyphenols, and Genetics: A Pilot Study in Overweight and Obese Adult Males to Determine Whether Black-Raspberry Consumption Affects Markers of Inflammation in Study Participants Fed a High-Fat, High-Calorie Challenge Meal
Brief Title: Inflammation, Polyphenols, and Genetics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Joseph Kitzmiller, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: OSU 2011H0394
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Overweight; Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blackraspberry slurry, washout, water (Experimental): Blackraspberry slurry daily x 5 days, 2 day washout, 8 oz. water daily x 5 days
  Interventions: Dietary Supplement: Blackraspberry Slurry
- Water, washout, Blackraspberry slurry (Experimental): 8 oz. water daily x 5 days, 2 day washout, Blackraspberry slurry daily x 5 days
  Interventions: Dietary Supplement: Blackraspberry Slurry

INTERVENTIONS:
Dietary Supplement: Blackraspberry Slurry — Blackraspberry slurry is 45 g blackraspberry powder mixed in 8oz. water. This is equivalent to 450 g fresh black raspberries.

SUMMARY:
Pilot study to determine whether daily consumption of blackraspberry powder (high in polyphenols) can reduce markers of inflammation and to determine whether genetics influence baseline levels of inflammatory markers as well as individual's response to polyphenols. A total of 10 males participated in this cross-over study.

DETAILED DESCRIPTION:
A high-fat, high-calorie challenge meal is administered to induce an inflammatory response in overweight and obese adult males. Serum levels of CRP, TNF-alpha, and IL-6 are measured prior to the challenge meal and at various times (1,2,4,8, and 12 hours) after the challenge meal. The challenge meal is given once without intervention and once after 5 daily doses of concentrated black-raspberry powder mixed in water.

ELIGIBILITY:
Inclusion Criteria:

* adult males over 55 years of age
* overweight or obese

Exclusion Criteria:

* history of adverse reaction to berries or berry products
* history of adverse reaction to high-fat, high-calorie challenge meal
* significant liver or renal insufficiency
* significant cognitive impairment

Min Age: 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Kitzmiller, MD PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Univesity, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sardo CL, Kitzmiller JP, Apseloff G, Harris RB, Roe DJ, Stoner GD, Jacobs ET. An Open-Label Randomized Crossover Trial of Lyophilized Black Raspberries on Postprandial Inflammation in Older Overweight Males: A Pilot Study. Am J Ther. 2016 Jan-Feb;23(1):e86-91. doi: 10.1097/MJT.0b013e3182a40bf8. PMID 23982695

RESULTS

PARTICIPANT FLOW:
Groups:
- Water First, Then Washout, Then Blackraspberry Slurry: 8 oz. water daily x 5 days, 2 day washout, Blackraspberry slurry daily x 5 days
- Blackraspberry Slurry First, Then Washout, Then Water: Blackraspberry slurry daily x 5 days, 2 day washout, 8 oz. water daily x 5 days
Period: First Intervention (6 Days)
Arm/Group | Water First, Then Washout, Then Blackraspberry Slurry | Blackraspberry Slurry First, Then Washout, Then Water
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout (2 Days)
Arm/Group | Water First, Then Washout, Then Blackraspberry Slurry | Blackraspberry Slurry First, Then Washout, Then Water
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Intervention 2 (5 Days)
Arm/Group | Water First, Then Washout, Then Blackraspberry Slurry | Blackraspberry Slurry First, Then Washout, Then Water
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: older obese and overweight males
Groups:
- Black-raspberry Powder: Black-raspberry powder: Black-raspberry powder (45g) equivalent to about 450 g fresh black raspberries
- No Intervention: Water without lypholized black raspberry powder
- Total: Total of all reporting groups
Arm/Group | Black-raspberry Powder | No Intervention | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.9) | 64.7 (6.9) | 64.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Serum IL-6
Description: Area Under the time-concentration Curve (AUC) of IL-6
Time Frame: acute (0-12 hours) after inflammation-causing challenge meal
Measure: Mean (95% Confidence Interval); unit: (pg*hr)/mL
Groups:
- Water: Water without lypholized black raspberry powder
- Blackraspberry Slurry: Blackraspberry slurry: Black-raspberry powder (45g) equivalent to about 450 g fresh black raspberries mixed with 8 oz water
Arm/Group | Water | Blackraspberry Slurry
Number analyzed (Participants) | 10 | 10
(pg*hr)/mL | 42.4 [24.5 to 60.3] | 34.3 [24.5 to 41.9]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Black-raspberry Slurry, Washout, Water; Water, Washout, Black-raspberry Slurry: Black-raspberry Slurry: Black-raspberry powder (45g) equivalent to about 450 g fresh black raspberries.
Arm/Group | Black-raspberry Slurry, Washout, Water | Water, Washout, Black-raspberry Slurry
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No